CLINICAL TRIAL: NCT02943850
Title: Human Neural Progenitor Cells Secreting Glial Cell Line-Derived Neurotrophic Factor (CNS10-NPC-GDNF) for the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: CNS10-NPC-GDNF for the Treatment of ALS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Principal Investigator, Robert H. Baloh, Director of Neuromuscular Medicine, ALS Program Director, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00042350
Record Dates: First submitted 2016-10-20; First posted 2016-10-25 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: stem cells; growth factor; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Stem cell implantation (Experimental): Subjects meeting all Eligibility Criteria and providing Informed Consent will be enrolled in one of two sequential dosing groups (Group A and B). Subjects will be treated sequentially with a minimum of one month interval between surgeries for the first three subjects in each dosing cohort. The remaining subjects in the cohort will be treated with a minimum interval of at least one week between surgeries. There will be 9 subjects in each group. No control group is included. All patients will received unilateral lumbar spinal cord injections of CNS10-NPC-GDNF cells.
  Interventions: Biological: Stem cell (HPC) implantation; Device: Stereotactic surgical device

INTERVENTIONS:
Biological: Stem cell (HPC) implantation — All patients will received unilateral lumbar spinal cord injections of CNS10-NPC-GDNF cells.
Device: Stereotactic surgical device — A newly developed stereotactic frame is being evaluated as a part of this trial

SUMMARY:
The investigator is examining the safety of transplanting cells that have been engineered to produce a growth factor into the spinal cord of patients with Amyotrophic Lateral Sclerosis (ALS). The cells are called neural progenitor cells, which are a type of stem cell that can become several different types of cells in the nervous system. These cells have been derived to specifically become astrocytes, which is a type of neuronal cell. The growth factor is called glial cell line-derived neurotrophic factor, or GDNF. GDNF is a protein that promotes the survival of many types of neuronal cells. Therefore, the cells are called "CNS10-NPC-GDNF." The investigational treatment has been tested in animals, but it has not yet been tested in people. In this study, we want to learn if CNS10-NPC-GDNF cells are safe to transplant into the spinal cords of people.

DETAILED DESCRIPTION:
This study will be the first to use a genetically modified progenitor cells to treat a neurodegenerative disease. This is a Phase 1/2a, single-center, blinded (as to side of injection), safety study of two escalating doses of human neural progenitor cells expressing GDNF (CNS10-NPC-GDNF) delivered unilaterally to the lumbar region in ALS subjects with moderate leg involvement.

Subjects meeting all Eligibility Criteria and providing Informed Consent will be enrolled in one of two sequential dosing groups. Subjects will be treated sequentially with a minimum of one month interval between surgeries for the first three subjects in each dosing cohort. The remaining subjects in the cohort will be treated with a minimum interval of at least two weeks between surgeries.

Specific aims:

Safety, as evaluated by:

* Adverse Events and Serious Adverse Events
* Clinical laboratory assessments, as clinically indicated (hematology, chemistry, immunology)

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of ALS (Lab-supported Probable, Probable or Definite EI Escorial Criteria)
2. Duration of symptoms ≤ 36 months
3. Progressive weakness in lower extremities, with EMG supported evidence of denervation in both lower extremities.
4. Forced Vital Capacity >60% of predicted normal in supine.
5. Male/Female; Age: 18 and older
6. Able to provide Informed Consent
7. Be geographically accessible to the study site and able to travel to study site for required visits
8. Have caregiver to assist in the transportation and care required by participation in the study
9. Not taking riluzole or on a stable dose for ≥ 30 days
10. For women of child bearing capacity, negative pregnancy test prior to surgery
11. Medically able to undergo thoracolumbar laminectomy or laminoplasty as determined by the site PI and Neurosurgeon
12. Medically able to tolerate the immunosuppression regimen as determined by the site PI

Exclusion Criteria:

1. Using invasive ventilatory assistance
2. Diagnosis of another active or unstable medical illness that may interfere with study participation at discretion of PI
3. Presence of any of the following conditions:

   1. Current drug or alcohol abuse
   2. Any known immunodeficiency syndrome
   3. Unstable medical condition
   4. Unstable psychiatric illness including psychosis and untreated major depression within 90 days of screening
4. Persons of child bearing capacity not willing to practice birth control
5. Receiving any investigational device/biologic/drug in past 30 days or any previous exposure to stem cell therapy
6. Any condition in the lower extremities which precludes serial strength testing
7. Any condition that the Neurosurgeon feels may pose complications for the surgery
8. Any condition or ALS disease phenotype that the site PI feels may interfere with participation in the study or in the interpretation of study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Safety evaluated by Adverse Events and Serious Adverse Events, post-operative MRI, and clinical laboratory assessments | Patients will be followed postoperatively for 12 months
  Safety, as evaluated by:
  * Adverse Events and Serious Adverse Events
  * Post-op MRI
  * Clinical laboratory assessments, as clinically indicated (hematology, chemistry, immunology)

SECONDARY OUTCOMES:
Compound Motor Action Potential (CMAP) | CMAP will be performed 7 times over 15 months
  Compound Motor Action Potential - CMAP (Tibialis anterior)
Force Generation via ATLIS testing | ATLIS testing will be performed 7 times over 15 months
  Lower extremity Force Generation via ATLIS testing
Quantitative Muscle MRI | Muscle MRI will be performed 6 times over 15 months
  Quantitative Muscle MRI of bilateral lower extremities
Electrical Impedance Myography (EIM) | EIM will be performed 7 times over 15 months
  Lower Extremity Electrical Impedance Myography (EIM)
Assessment of glial cell line derived neurotrophic factor (GDNF) in the cerebral spianl fluid (CSF) | CSF will be collected at 3 time points over 12 months
  Assessment of GDNF in the CSF

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Baloh, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baloh RH, Johnson JP, Avalos P, Allred P, Svendsen S, Gowing G, Roxas K, Wu A, Donahue B, Osborne S, Lawless G, Shelley B, Wheeler K, Prina C, Fine D, Kendra-Romito T, Stokes H, Manoukian V, Muthukumaran A, Garcia L, Banuelos MG, Godoy M, Bresee C, Yu H, Drazin D, Ross L, Naruse R, Babu H, Macklin EA, Vo A, Elsayegh A, Tourtellotte W, Maya M, Burford M, Diaz F, Patil CG, Lewis RA, Svendsen CN. Transplantation of human neural progenitor cells secreting GDNF into the spinal cord of patients with ALS: a phase 1/2a trial. Nat Med. 2022 Sep;28(9):1813-1822. doi: 10.1038/s41591-022-01956-3. Epub 2022 Sep 5. PMID 36064599